CLINICAL TRIAL: NCT06806696
Title: SARS-COV-2 VARIANTS' EFFECT ON PREGNANCY AND LONG-TERM OUTCOMES AMONG PREGNANT WOMEN AND THEIR NEWBORNS IN ESTONIA
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Irja Lutsar, Professor of Medical Microbiology, University of Tartu
Other Study IDs: 382/M-8
Record Dates: First submitted 2025-01-22; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; COVID-19; Post-COVID / Long-COVID; Newborn Health; Miscarriages
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with COVID-19 and their offspring: Pregnant women who were diagnosed with COVID-19 during the study period, along with their offspring
  Interventions: Other: COVID-19 infection
- Pregnant women who did not have COVID-19 and their offspring: Pregnant women who did not have COVID-19 during pregnancy, along with their offspring

INTERVENTIONS:
Other: COVID-19 infection — COVID-19 diagnosis in the health database
  Groups: Pregnant women with COVID-19 and their offspring

SUMMARY:
The main aim of the study is to describe the possible impacts of SARS-CoV-2 and its various genotypes on pregnancy and long-term outcomes among pregnant women and their newborns in Estonia.

DETAILED DESCRIPTION:
All the pregnant women in Estonia who conceived and gave birth between February 27, 2020, and March 1, 2023 were included in the study. Pregnant women will be divided into 2 groups: 1. pregnant women who were diagnosed with COVID-19 during the study period, along with their newborns; 2. control group: pregnant women who did not have COVID-19 during pregnancy, along with their newborns. The following data is collected for each subject: prior vaccination, previous COVID-19 infection, underlying diseases/conditions, hospitalization, need for intensive care, need for mechanical ventilation and/or oxygen therapy, death cases, post-COVID-19 symptoms, pregnancy course and outcomes, possible virus transmission from mother to child, and the newborn's condition or accompanying health issues

ELIGIBILITY:
Inclusion Criteria:

* pregnancy (conceived and gave birth between February 27, 2020, and March 1, 2023) with COVID-19 or without and their newborns

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the pregnant Estonian women who conceived and gave birth between February 27, 2020, and March 1, 2023
Sampling Method: Probability Sample
Enrollment: 60739 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 incidence | From enrollment to March 2023
Post-COVID condition incidence | From enrollment to March 2023
Chronic diseases incidence | From enrollment to March 2023
Newborn condition | From enrollment to March 2023
  Apgar scores at birth
Mortality | From enrollment to March 2023
Hospitalization rate due to COVID-19 | From enrollment to March 2023
Pregnancy complications incidence | From enrollment to March 2023

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No
The IPD collected throughout this trial will not be shared due to data protection laws.